CLINICAL TRIAL: NCT01370850
Title: Clinical Validation Study of RTVue Features
Status: Completed | Type: Observational
Sponsor: Optovue (Industry)
Responsible Party: Mike Sinai, PhD / Director of Clinical Affairs, Optovue
Other Study IDs: RTVue Validation Study
Record Dates: First submitted 2011-04-28; First posted 2011-06-10 (Estimated); Last update posted 2011-06-10 (Estimated); Status verified 2011-06

CONDITIONS: Healthy; Glaucoma
Keywords: Retina pathology
MeSH Terms: conditions — Glaucoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Normal: Normal results from the clinical exam and free of ocular pathology.
- Glaucoma: Clinical exam results consistent with glaucoma; visual field defects consistent with glaucoma and/or structural damage consistent with glaucoma.
- Retina: Clinical exam results consistent with retina pathology.

SUMMARY:
To perform a clinical validation study of RTVue features in volunteers with various ocular pathology or no ocular pathology.

DETAILED DESCRIPTION:
Clinical validation study of RTVue features in volunteers with various ocular pathology or no ocular pathology. Subjects to undergo a clinical exam and OCT scanning.

ELIGIBILITY:
Inclusion Criteria:

* Normal subjects will have normal results from the clinical exam and be free of ocular pathology.
* Glaucoma patients will have clinical exam results consistent with glaucoma; they will have visual field defects consistent with glaucoma and/or structural damage consistent with glaucoma.
* Retina patients will have clinical exam results consistent with retina pathology.

Exclusion Criteria:

* Normal subjects will be free of any ocular pathology.
* Glaucoma patients will be free of any ocular pathology except glaucoma.
* Retina patients will be free of any ocular pathology except any type of retina pathology.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Volunteers with various ocular pathology or no ocular pathology
Sampling Method: Non-Probability Sample
Enrollment: 53 (Actual)
Dates: Start 2011-03; Primary Completion 2011-04 (Actual); Study Completion 2011-04 (Actual)

PRIMARY OUTCOMES:
Retina measurement | at time of study visit (day 1)

CONTACTS AND LOCATIONS:
Overall Officials: Mike Sinai, PhD, Study Director — Optovue
Locations (1):
- Pacific Eye Specialists, Daly City, California, United States